CLINICAL TRIAL: NCT03061201
Title: A PHASE 1/2, OPEN-LABEL, ADAPTIVE, DOSE-RANGING STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF SB-525 (PF-07055480) (RECOMBINANT AAV2/6 HUMAN FACTOR 8 GENE THERAPY) IN ADULT SUBJECTS WITH SEVERE HEMOPHILIA A
Brief Title: A Study of Recombinant AAV2/6 Human Factor 8 Gene Therapy SB-525 (PF-07055480) in Subjects With Severe Hemophilia A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-525-1603; C3731001 (Other: Alias Study Number)
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Dose selection based on safety and kinetics of circulating FVIII levels observed in previously dosed participants.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential dose escalation (Experimental): SB-525 (PF-07055480) is administered as a single infusion
  Interventions: Biological: SB-525 (PF-07055480)

INTERVENTIONS:
Biological: SB-525 (PF-07055480) — Single dose of investigational product SB-525 (PF-07055480)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and time-course profile of FVIII activity after dosing with SB-525 (PF-07055480)

DETAILED DESCRIPTION:
The proposed clinical study uses a recombinant adeno-associated virus 2/6 (AAV2/6) vector encoding the cDNA for the B-domain deleted human F8 (hF8). The secreted FVIII has the same amino acid sequence as approved recombinant anti hemophilic factors (Refacto® and Xyntha®). The SB-525 (PF-07055480) vector encodes a liver-specific promotor module and AAV2/6 exhibits liver tropism, thus providing the potential for long-term hepatic production of FVIII in hemophilia A subjects.

The constant production of FVIII after a single SB-525 (PF-07055480) administration may provide potential benefit in durable protection against bleeding and the complications thereof without lifelong repetitive IV factor replacement administration.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years of age
* Severe hemophilia A (past evidence of circulating FVIII activity of < 1% normal)
* Treated or exposed to FVIII concentrates or cryoprecipitate for at least 150 exposure days
* ≥12 bleeding episodes if receiving on-demand therapy over the preceding 12 months
* Agree to use double barrier contraceptive until at least 3 consecutive semen samples are negative for AAV 2/6 after SB-525 infusion

Exclusion Criteria:

* Presence of neutralizing antibodies
* Current inhibitor, or history of FVIII inhibitor (except for transient low titer inhibitor detected in childhood)
* History of hypersensitivity response to FVIII
* History of Hepatitis B or HIV-1/2 infection
* History of Hepatitis C, unless viral assays in two samples, collected at least 6 months apart, are negative
* Evidence of any bleeding disorder in addition to hemophilia A
* Markers of hepatic inflammation or overt or occult cirrhosis
* History of chronic renal disease or creatinine ≥ 1.5 mg/dL
* Presence of liver mass on magnetic resonance imaging (MRI), or, positive alpha fetoprotein
* Presence of > grade 2 liver fibrosis on elastography for subjects with history of treated Hepatitis C or suspicion of chronic liver disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope Medical Center, Duarte, California
  - Midtown Ambulatory Care Center, Sacramento, California
  - UC Davis Ambulatory Care Clinic, Sacramento, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC Davis CTSC Clinical Research Center, Sacramento, California
  - UC Davis Hemophilia Treatment Center, Sacramento, California
  - UC Davis Investigational Drug Services Pharmacy, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - University of California, San Francisco - Investigational Drug Service (IDS) Pharmacy, San Francisco, California
  - University of California, San Francisco - Outpatient Hematology Clinic, San Francisco, California
  - University of California, San Francisco -Moffitt Hospital, San Francisco, California
  - University Of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - UPMC Montefiore Clinical and Translational Research Center, Pittsburgh, Pennsylvania
  - UPMC, Investigational Drug Service, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center Clinical Research Center, Nashville, Tennessee
  - Vanderbilt Hemostasis Treatment Clinic, Nashville, Tennessee
  - Vanderbilt Hemostasis-Thrombosis Clinic, Nashville, Tennessee
  - Washington Institute for Coagulation, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Leavitt AD, Konkle BA, Stine KC, Visweshwar N, Harrington TJ, Giermasz A, Arkin S, Fang A, Plonski F, Yver A, Ganne F, Agathon D, Resa MLA, Tseng LJ, Di Russo G, Cockroft BM, Cao L, Rupon J. Giroctocogene fitelparvovec gene therapy for severe hemophilia A: 104-week analysis of the phase 1/2 Alta study. Blood. 2024 Feb 29;143(9):796-806. doi: 10.1182/blood.2022018971. PMID 37871576
- [Derived] Cao L, Ledeboer A, Pan Y, Lu Y, Meyer K. Clinical enrollment assay to detect preexisting neutralizing antibodies to AAV6 with demonstrated transgene expression in gene therapy trials. Gene Ther. 2023 Feb;30(1-2):150-159. doi: 10.1038/s41434-022-00353-2. Epub 2022 Jul 1. PMID 35778500
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SB-525-1603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with severe hemophilia A were enrolled in this study and received single infusion of SB-525/ PF-07055480. Participants were followed up for maximum of 5 years post-infusion.
Groups:
- Cohort 1: PF-07055480 9*10^11 vg/kg: Participants received a single intravenous infusion of PF-07055480 9.0*10^11 vector genomes per kilogram (vg/kg) on Day 1.
- Cohort 2: PF-07055480 2*10^12 vg/kg: Participants received a single intravenous infusion of PF-07055480 2.0*10^12 vg/kg on Day 1.
- Cohort 3: PF-07055480 1*10^13 vg/kg: Participants received a single intravenous infusion of PF-07055480 1.0*10^13 vg/kg on Day 1.
- Cohort 4: PF-07055480 3*10^13 vg/kg: Participants received a single intravenous infusion of PF-07055480 3.0*10^13 vg/kg on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Started | 2 | 2 | 2 | 5
Completed | 1 | 1 | 2 | 4
Not Completed | 1 | 1 | 0 | 1
Not completed — Participants Terminated at Month 36 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: PF-07055480 9*10^11 vg/kg: Participants received a single intravenous infusion of PF-07055480 9.0*10^11 vg/kg on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.50 (9.192) | 35.50 (16.263) | 32.00 (1.414) | 26.80 (6.301) | 30 (7.937)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 2 | 2 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race is reported.
  Participants
    Race: Asian | 0 | 1 | 0 | 0 | 1
    Race: White | 2 | 1 | 2 | 4 | 9
    Race: Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the criteria as follows: death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly/birth defect and other situations per protocol. AEs included both SAEs and all non-SAEs.
Time Frame: From Baseline (1 week prior to infusion) up to 5 years post-infusion (approximately 5 Years)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Participants
  Participants With AEs | 2 | 2 | 2 | 5
  Participants With SAEs | 0 | 2 | 0 | 1

2. Primary Outcome: Central FVIII Activity Levels by Chromogenic Assay at Year 1 (Week 52)
Description: FVIII activity levels were assessed using chromogenic and one-stage clotting assay and which were analyzed in the central laboratory. In this outcome measure results by chromogenic assay are reported.
Time Frame: At Year 1 (Week 52)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. For Cohort 1, both participants resumed prophylaxis regimen prior to Week 52, and were excluded from analysis as pre-specified in the Statistical Analysis Plan (SAP).
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 2 | 1 | 4
Percentage of Normal |  | 0.90 (0.000) | 11.90 | 42.60 (53.473)

3. Primary Outcome: Central FVIII Activity Levels by Chromogenic Assay at Year 2 (Week 104)
Description: as for outcome 2
Time Frame: At Year 2 (Week 104)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. For Cohort 1, both participants resumed prophylaxis regimen prior to Week 52, and were excluded from analysis as pre-specified in the SAP.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 5
Percentage of Normal |  | 19.30 | 8.25 | 25.44 (27.532)

4. Primary Outcome: Central FVIII Activity Levels by Chromogenic Assay at Year 3 (Week 156)
Description: as for outcome 2
Time Frame: At Year 3 (Week 156)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 5
Percentage of Normal |  | 0.90 | 4.40 | 25.46 (36.998)

5. Primary Outcome: Central FVIII Activity Levels by Chromogenic Assay at Year 4 (Week 208)
Description: as for outcome 2
Time Frame: At Year 4 (Week 208)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 4
Percentage of Normal |  | 0.90 | 3.20 | 26.55 (42.489)

6. Primary Outcome: Central FVIII Activity Levels by Chromogenic Assay at Year 5 (Week 260)
Description: as for outcome 2
Time Frame: At Year 5 (Week 260)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 4
Percentage of Normal |  | 0.90 | 3.30 | 23.55 (36.270)

7. Primary Outcome: Central FVIII Activity Levels by One-Stage Clotting Assay at Year 1 (Week 52)
Description: FVIII activity levels were assessed using chromogenic and one-stage clotting assay and which were analyzed in the central laboratory. In this outcome measure results by one-stage clotting assay are reported.
Time Frame: At Year 1 (Week 52)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 2 | 1 | 4
Percentage of Normal |  | 1.75 (1.202) | 19.90 | 66.37 (83.793)

8. Primary Outcome: Central FVIII Activity Levels by One-Stage Clotting Assay at Year 2 (Week 104)
Description: as for outcome 7
Time Frame: At Year 2 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 5
Percentage of Normal |  | 19.00 | 13.95 | 38.86 (36.738)

9. Primary Outcome: Central FVIII Activity Levels by One-Stage Clotting Assay at Year 3 (Week 156)
Description: as for outcome 7
Time Frame: At Year 3 (Week 156)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 5
Percentage of Normal |  | 3.30 | 5.70 | 40.52 (50.231)

10. Primary Outcome: Central FVIII Activity Levels by One-Stage Clotting Assay at Year 4 (Week 208)
Description: as for outcome 7
Time Frame: At Year 4 (Week 208)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 4
Percentage of Normal |  | 4.80 | 13.80 | 38.78 (53.790)

11. Primary Outcome: Central FVIII Activity Levels by One-Stage Clotting Assay at Year 5 (Week 260)
Description: as for outcome 7
Time Frame: At Year 5 (Week 260)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 4
Percentage of Normal |  | 4.00 | 6.10 | 41.00 (56.749)

12. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by Chromogenic Assay at Yearly Interval 1 (Week 9 Through Week 53)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by chromogenic assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 1 included assessments from Week 9 through Week 53). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 1 (Week 9 through Week 53)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. As pre-specified in planned analysis in the statistical analysis plan (SAP) of the study, this outcome measure was to be assessed only in Cohort 4.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 67.89 (46.585)

13. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by Chromogenic Assay at Yearly Interval 2 (Week 54 Through Week 108)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by chromogenic assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 2 included assessments from Week 54 through Week 108). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 2 (Week 54 through Week 108)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. As pre-specified in planned analysis in the SAP of the study, this outcome measure was to be assessed only in Cohort 4.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 40.38 (41.498)

14. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by Chromogenic Assay at Yearly Interval 3 (Week 109 Through Week 160)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by chromogenic assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 3 included assessments from Week 109 through Week 160). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 3 (Week 109 through Week 160)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 27.66 (41.589)

15. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by Chromogenic Assay at Yearly Interval 4 (Week 161 Through Week 212)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by chromogenic assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 4 included assessments from Week 161 through Week 212). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 4 (Week 161 through Week 212)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. As pre-specified in planned analysis in the SAP of the study, this outcome measure was to be assessed only in Cohort 4. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 4
Percentage of Normal | 24.31 (34.640)

16. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by Chromogenic Assay at Yearly Interval 5 (Week 213 Through Week 264)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by chromogenic assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 5 included assessments from Week 213 through Week 264). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 5 (Week 213 through Week 264)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 4
Percentage of Normal | 24.87 (39.509)

17. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by One-Stage Clotting Assay at Yearly Interval 1 (Week 9 Through Week 53)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by one-stage clotting assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 1 included assessments from Week 9 through Week 53). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 1 (Week 9 through Week 53)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 107.44 (72.860)

18. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by One-Stage Clotting Assay at Yearly Interval 2 (Week 54 Through Week 108)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by one-stage clotting assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 2 included assessments from Week 54 through Week 108). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 2 (Week 54 through Week 108)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 58.55 (56.752)

19. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by One-Stage Clotting Assay at Yearly Interval 3 (Week 109 Through Week 160)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by one-stage clotting assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 3 included assessments from Week 109 through Week 160). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 3 (Week 109 through Week 160)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 5
Percentage of Normal | 43.95 (57.466)

20. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by One-Stage Clotting Assay at Yearly Interval 4 (Week 161 Through Week 212)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by one-stage clotting assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 4 included assessments from Week 161 through Week 212). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 4 (Week 161 through Week 212)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 4
Percentage of Normal | 39.60 (51.623)

21. Primary Outcome: Geometric Mean of Central FVIII Activity Levels for Cohort 4 by One-Stage Clotting Assay at Yearly Interval 5 (Week 213 Through Week 264)
Description: FVIII activity levels were analyzed in the central laboratory using chromogenic and one-stage clotting assay. In this outcome measure FVIII activity levels were assessed by one-stage clotting assay. As pre-specified, for each participant geometric mean of central FVIII activity levels was calculated of all eligible FVIII activity measurements for each yearly interval (for this outcome measure: Yearly Interval 5 included assessments from Week 213 through Week 264). Following this mean and standard deviation as summary statistics across all evaluable participants was calculated and is reported as data for this outcome measure.
Time Frame: Year 5 (Week 213 through Week 264)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 4
Percentage of Normal | 38.62 (51.844)

22. Secondary Outcome: Total Annualized Bleeding Rate (ABR)
Description: Total ABR included both treated and untreated bleeding episodes. In this outcome measure total ABR for pre-screening and post-infusion are reported. Pre-screening total ABR was based on the total number of reported bleeding episodes during 12 months prior to screening visit as reported on CRF's Hemophilia A History page. Screening was 2 months before baseline. Post- infusion total ABR = number of all bleeding episodes starting 3 weeks after investigational product/ PF-07055480 (IP) infusion up to date of day before start of prophylaxis (or date of data cut or conclusion date)/ observation period in years, where observation period in years = date of day before start of prophylaxis or date of data cut or conclusion date - 3 weeks after date of IP infusion + 1)/365.25. For a participant who did not start prophylaxis the data cut date or conclusion date is used.
Time Frame: Pre-screening period: 12 months prior to screening; Post-infusion period: 3 weeks post-infusion up to date of day before start of prophylaxis or date of data cut or conclusion date, whichever was earlier (maximum up to 5 years)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Bleeds per year
  Pre-screening total ABR | 3.50 (0.707) | 14.00 (16.971) | 1.50 (2.121) | 8.80 (8.319)
  Post infusion total ABR -until prophylaxis is resumed | 7.93 (3.139) | 3.07 (2.898) | 3.24 (4.586) | 1.53 (3.235)

23. Secondary Outcome: Total ABR by Severity
Description: Total ABR include both treated and untreated bleeding episodes. In this outcome measure total ABR by severity for post-infusion period is reported. Severity was categorized as mild, moderate and severe. Post- infusion total ABR = number of all bleeding episodes starting 3 weeks after IP infusion up to date of day before start of prophylaxis (or date of data cut or conclusion date)/ observation period in years, where observation period in years = date of day before start of prophylaxis or date of data cut or conclusion date - 3 weeks after date of IP infusion + 1)/365.25. For a participant who did not start prophylaxis the data cut date or conclusion date is used.
Time Frame: Post-infusion period: 3 weeks post-infusion up to date of day before start of prophylaxis or date of data cut or conclusion date, whichever was earlier (maximum up to 5 years)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Bleeds per year
  Mild | 7.93 (3.139) | 0.87 (0.081) | 0.17 (0.241) | 1.22 (2.725)
  Moderate | 0.00 (0.000) | 1.73 (2.159) | 3.07 (4.345) | 0.31 (0.528)
  Severe | 0.00 (0.000) | 0.47 (0.658) | 0.00 (0.000) | 0.00 (0.000)

24. Secondary Outcome: Annualized Infusion Rate (AIR)
Description: AIR was calculated and reported for pre-infusion and post-infusion. AIR for pre-infusion was calculated as, a) Excluding prophylaxis: number of FVIII replacement infusions for reasons other than prophylaxis prior to IP infusion/ ([date of IP infusion - date of screening] + 30)] *365.25, or b) number of FVIII replacement infusions for any reason prior to IP infusion/ ([date of IP infusion - date of screening] + 30)] *365.25. Screening was 2 months before baseline and baseline was approximately 1-week prior to IP infusion. AIR for post- infusion was calculated as: number of FVIII replacement infusions started at 3 weeks after IP infusion up to date of data cut or conclusion date/ number of days in the observation period for the participant in years, where observation period in years = date of data cut or conclusion date - 3 weeks after date of IP infusion + 1)/365.25.
Time Frame: Pre-infusion period: 30 days before screening up to pre-infusion (approximately up to 3.23 months); post-infusion period: 3 weeks post-infusion up to up to date of data cut or conclusion date (maximum up to 5 years)
Population: Safety population included all participants enrolled in this study who received any portion of study intervention.
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Infusions per year
  Pre-infusion AIR (Excluding Prophylaxis) | 0.00 (0.00) | 2.10 (2.97) | 0.00 (0.00) | 1.62 (2.26)
  Pre-infusion AIR | 100.43 (2.74) | 81.15 (108.82) | 87.93 (118.73) | 120.86 (30.04)
  Post-infusion AIR | 58.95 (73.97) | 32.79 (25.32) | 29.03 (33.27) | 3.56 (7.55)

25. Secondary Outcome: Change From Baseline in the EuroQol, 5 Dimensions, 5 Levels (EQ-5D-5L) Index Score at Weeks 12, 24 and 52; Months 24, 36, 48 and 60
Description: EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group. It measures 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) of health on a 5-point scale. Each dimension had 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. EQ-5D-5L had 2 components: Index score and visual analogue scale (VAS). Index score was obtained, according to the health state defined by the 5 dimensions scores, from the Crosswalk Index value calculator and table lookup document under the target country population. A health state is defined by the combination of one level from each of the 5 dimensions. For this study, weights under the US population were used to obtain the Index score. Index score ranged between 0-1, where higher score indicates a better health state, and lower score indicate worse health state. Baseline was defined as the latest non-missing value before IP infusion.
Time Frame: Baseline; Weeks 12, 24, and 52; Months 24, 36, 48, and 60
Population: Safety population. Here, "Number Analyzed" =participants evaluable for specified timepoints. Participants from "Cohort 1: PF-07055480 9*10^11 vg/kg" and "Cohort 2: PF-07055480 2*10^12 vg/kg" did not attend the study visit or missed the EQ-5D-5L assessment at Months 24 and 60 and participants from "Cohort 3: PF-07055480 1*10^13 vg/kg" did not attend the study visit or missed the EQ-5D-5L assessment at Month 24; hence, no participants were analyzed for Cohorts 1, 2 and 3 at the mentioned visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Units on a scale
  Baseline | 0.902 (0.139) | 0.577 (0.254) | 0.922 (0.110) | 0.946 (0.122)
  Change at Week 12: number analyzed (Participants) | 2 | 1 | 2 | 5
  Change at Week 12 | 0.011 (0.016) | 0.244 | 0.078 (0.110) | 0.016 (0.035)
  Change at Week 24 | -0.033 (0.129) | 0.317 (0.103) | 0.078 (0.110) | -0.036 (0.080)
  Change at Week 52: number analyzed (Participants) | 2 | 2 | 1 | 5
  Change at Week 52 | -0.165 (0.266) | 0.294 (0.071) | 0.000 | -0.002 (0.004)
  Change at Month 24: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change at Month 24 |  |  |  | 0.000 (0.000)
  Change at Month 36: number analyzed (Participants) | 2 | 1 | 1 | 3
  Change at Month 36 | -0.099 (0.140) | 0.334 | -0.210 | 0.000 (0.000)
  Change at Month 48: number analyzed (Participants) | 1 | 1 | 1 | 3
  Change at Month 48 | -0.013 | 0.219 | -0.197 | 0.000 (0.000)
  Change at Month 60: number analyzed (Participants) | 0 | 0 | 2 | 4
  Change at Month 60 |  |  | -0.087 (0.047) | -0.053 (0.105)

26. Secondary Outcome: Change From Baseline in the EQ-5D-5L- VAS Score at Week 12, 24, 52 and Month 24, 36, 48, 60
Description: EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group. It measures 5 dimensions of health on a 5-point scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is assessed with 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. EQ-5D-5L had 2 components: Index score and VAS. EQ-5D-5L VAS: Participants were asked to indicate their current health status on a scale of 0 (worst health) to 100 (best imaginable health), higher scores signified better health status. Baseline was defined as the latest non-missing value before IP infusion.
Time Frame: Baseline; Weeks 12, 24, and 52; Months 24, 36, 48, and 60
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Units on a scale
  Baseline | 75.0 (7.07) | 73.5 (9.19) | 80.0 (14.14) | 92.6 (10.67)
  Change at Week 12: number analyzed (Participants) | 2 | 1 | 2 | 5
  Change at Week 12 | 4.5 (6.36) | 10.0 | 5.0 (21.21) | -0.4 (5.32)
  Change at Week 24 | 10.0 (7.07) | 15.0 (0.00) | 19.5 (14.85) | -3.0 (7.52)
  Change at Week 52: number analyzed (Participants) | 2 | 2 | 1 | 5
  Change at Week 52 | -1.0 (12.73) | 16.0 (1.41) | -10.0 | -4.2 (6.57)
  Change at Month 24: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change at Month 24 |  |  |  | -4.0 (5.66)
  Change at Month 36: number analyzed (Participants) | 2 | 1 | 1 | 3
  Change at Month 36 | 0.0 (0.0) | 8.0 | 0.0 | -0.7 (9.02)
  Change at Month 48: number analyzed (Participants) | 1 | 1 | 1 | 3
  Change at Month 48 | 0.0 | 10.0 | 0.0 | -3.0 (3.00)
  Change at Month 60: number analyzed (Participants) | 0 | 0 | 2 | 4
  Change at Month 60 |  |  | 4.5 (6.36) | -1.3 (9.07)

27. Secondary Outcome: Number of Participants With Positive FVIII Inhibitor Levels During the Study
Description: Positive FVIII inhibitor was assessed using central laboratory using Nijmegen method of the Bethesda assay in an individual with no prior history of FVIII inhibitor. Inhibitor assay results >0.6 Bethesda units (BU) were considered as positive. Positive results at any timepoint were considered, even if subsequent inhibitor assessment was negative.
Time Frame: Baseline (one week prior to IP infusion) up to 5 years post-infusion
Population: Safety population included all participants enrolled in this study who received any portion of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Participants | 1 | 0 | 0 | 0

28. Secondary Outcome: Peak Value of AAV2/6 (Adeno-associated Vector 2/6) Deoxyribonucleic Acid (DNA) in Plasma, Saliva, Semen, Stool and Urine
Description: Peak (maximum) AAV2/6 vector DNA concentration (vg/mL) in plasma, saliva, semen, stool and urine were analyzed with quantitative real-time polymerase chain reaction (PCR). Participants must achieve 3 consecutive negative results for analysis for each sample.
Time Frame: All samples: Baseline, Day 7, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and every month after Week 52 until Month 60 until 3 consecutive negative samples are obtained on a sample-type basis; additional for plasma at 12 hours post-infusion
Population: Safety population included all participants enrolled in this study who received any portion of study intervention. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Vector genome per milliliter (vg/mL)
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Vector genome per milliliter (vg/mL)
  Plasma | 25680000 (26620000) | 292600000 (383900000) | 1787000000 (1390000000) | 3442000000 (2809000000)
  Saliva | 44550 (21710) | 159500 (89870) | 1555000 (417200) | 6972000 (5158000)
  Semen: number analyzed (Participants) | 1 | 1 | 2 | 5
  Semen | 14600 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 36500 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 145500 (4950) | 99780 (151900)
  Stool: number analyzed (Participants) | 2 | 0 | 2 | 5
  Stool | 604 (407.3) |  | 2490 (2461) | 2277 (2814)
  Urine: number analyzed (Participants) | 0 | 0 | 0 | 3
  Urine |  |  |  | 9697 (6166)

29. Secondary Outcome: Time to Peak Value of AAV2/6 Vector DNA in Plasma, Saliva, Semen, Stool and Urine
Description: Time to peak (maximum) AAV2/6 vector DNA concentration (vg/mL) in plasma, saliva, urine, stool and semen were analyzed with quantitative real-time PCR. Participants must achieve 3 consecutive negative results for analysis for each sample; where negative suggests values under the limit of detection.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Days
  Plasma | 1.5 (0.71) | 1.0 (0.00) | 1.0 (0.00) | 1.4 (0.55)
  Saliva | 11.5 (4.95) | 7.5 (0.71) | 12.0 (4.24) | 11.8 (3.96)
  Semen: number analyzed (Participants) | 1 | 1 | 2 | 5
  Semen | 8.0 | 15.0 | 11.0 (4.24) | 14.4 (8.99)
  Stool: number analyzed (Participants) | 2 | 0 | 2 | 5
  Stool | 8.0 (0.00) |  | 7.5 (0.71) | 17.0 (10.32)
  Urine: number analyzed (Participants) | 0 | 0 | 0 | 3
  Urine |  |  |  | 9.7 (3.79)

30. Secondary Outcome: Time to Undetectable (Negative) Value of AAV2/6 Vector DNA in Plasma, Saliva, Semen, Stool and Urine
Description: Time to undetectable (negative) value of AAV2/6 vector DNA concentration (vg/mL) in plasma, saliva, urine, stool and semen were analyzed with quantitative real-time PCR. Time to undetectable is defined as the number of days from IP infusion until the first of 3 consecutive specimens under the limit of detection (negative).
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Days
  Plasma: number analyzed (Participants) | 2 | 2 | 2 | 3
  Plasma | 22.0 (8.49) | 15.0 (0.00) | 56.5 (0.71) | 84.7 (47.92)
  Saliva: number analyzed (Participants) | 2 | 2 | 2 | 4
  Saliva | 28.5 (0.71) | 29.0 (0.00) | 56.5 (0.71) | 60.5 (17.62)
  Semen: number analyzed (Participants) | 2 | 1 | 2 | 5
  Semen | 18.0 (14.14) | 15.0 | 42.0 (18.38) | 42.2 (27.51)
  Stool: number analyzed (Participants) | 1 | 1 | 2 | 5
  Stool | 15.0 | 15.0 | 42.0 (18.38) | 72.6 (62.10)
  Urine | 8.0 (0.00) | 7.5 (0.71) | 8.5 (0.71) | 14.8 (8.17)

31. Secondary Outcome: Time to Last of 3 Consecutive Negative Values of AAV2/6 Vector DNA in Plasma, Saliva, Semen, Stool and Urine
Description: Time to last of 3 consecutive negative value of AAV2/6 vector DNA concentration (vg/mL) in plasma, saliva, urine, stool and semen were analyzed with quantitative real-time PCR.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Days
  Plasma: number analyzed (Participants) | 2 | 2 | 2 | 3
  Plasma | 71.0 (19.80) | 57.0 (0.00) | 113.5 (0.71) | 166.7 (92.95)
  Saliva: number analyzed (Participants) | 2 | 2 | 2 | 4
  Saliva | 85.0 (0.00) | 84.5 (0.71) | 113.5 (0.71) | 105.3 (27.60)
  Semen: number analyzed (Participants) | 2 | 1 | 2 | 5
  Semen | 55.5 (40.31) | 57.0 | 115.5 (43.13) | 95.4 (31.41)
  Stool: number analyzed (Participants) | 1 | 1 | 2 | 5
  Stool | 56.0 | 84.0 | 115.5 (43.13) | 185.6 (164.77)
  Urine | 28.5 (0.71) | 29.0 (0.00) | 28.5 (0.71) | 45.4 (14.99)

32. Secondary Outcome: Time to Last Positive Value Prior to First of 3 Consecutive Negatives of AAV2/6 Vector DNA in Plasma, Saliva, Semen, Stool and Urine
Description: Time to last positive value prior to first of 3 consecutive negatives of AAV2/6 vector DNA concentration (vg/mL) in plasma, saliva, urine, stool and semen were analyzed with quantitative real-time PCR, where positive suggests values above the limit of detection.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5
Days
  Plasma: number analyzed (Participants) | 2 | 2 | 2 | 3
  Plasma | 11.5 (4.95) | 7.5 (0.71) | 28.5 (0.71) | 47.3 (31.75)
  Saliva: number analyzed (Participants) | 2 | 2 | 2 | 4
  Saliva | 15.5 (0.71) | 15.0 (0.00) | 28.5 (0.71) | 35.5 (14.34)
  Semen: number analyzed (Participants) | 1 | 0 | 2 | 5
  Semen | 15.0 |  | 21.5 (9.19) | 18.6 (9.56)
  Stool: number analyzed (Participants) | 1 | 0 | 2 | 5
  Stool | 8.0 |  | 21.5 (9.19) | 21.4 (9.66)
  Urine: number analyzed (Participants) | 0 | 0 | 0 | 3
  Urine |  |  |  | 9.7 (3.79)

ADVERSE EVENTS:
Time Frame: From Baseline (1 week prior to infusion) up to 5 years post-infusion (approximately 5 Years)
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as SAE in one participant and as non-SAE in another participant, or one participant may have experienced both a serious and non-SAE event during the study. Safety population included all participants who enrolled in this study who received any portion of study intervention.
Arm/Group | Cohort 1: PF-07055480 9*10^11 vg/kg | Cohort 2: PF-07055480 2*10^12 vg/kg | Cohort 3: PF-07055480 1*10^13 vg/kg | Cohort 4: PF-07055480 3*10^13 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-07055480 9*10^11 vg/kg (N=2) | Cohort 2: PF-07055480 2*10^12 vg/kg (N=2) | Cohort 3: PF-07055480 1*10^13 vg/kg (N=2) | Cohort 4: PF-07055480 3*10^13 vg/kg (N=5)
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Perineal cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-07055480 9*10^11 vg/kg (N=2) | Cohort 2: PF-07055480 2*10^12 vg/kg (N=2) | Cohort 3: PF-07055480 1*10^13 vg/kg (N=2) | Cohort 4: PF-07055480 3*10^13 vg/kg (N=5)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 3
Coagulation factor VIII level increased (Investigations) | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Any untoward clinically significant changes from pre vector dosing identified on physical examinations, clinical laboratory assessments, immune parameters, liver imaging, vital signs, Electrocardiogram during the during study were captured as AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT03061201/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT03061201/SAP_001.pdf